CLINICAL TRIAL: NCT04713605
Title: Cerebral Blood Flow in Neonates During Major Cardiac- and Non-cardiac Surgery
Brief Title: Cerebral Blood Flow in Neonates During Major Cardiac Surgery.
Acronym: FLOWER
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Kim van Loon, Principle investigator, UMC Utrecht
Other Study IDs: NL76532.041.21
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Hypoperfusion in Newborn With Congenital Heart Disease
Keywords: TCD; hypoperfusion; critical closing pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Critical closing pressure detection — Observational study that determines the critical closing pressure (CrCP) of the brain by comparison of the cerebral blood flow velocity (measured by TCD) and invasive blood pressure measurement (IABP)

SUMMARY:
Rationale: During cardiac surgery, neonates are at high risk of cerebral damage: 36-78% will have new cerebral lesions after surgery. Adequate cerebral perfusion (CBF) is mandatory to prevent postoperative brain damage and neurobehavioral outcomes. For CBF, the systemic blood pressure should be managed above the brain's critical closing pressure (CrCP), and preferably above the lower limit of autoregulation (LLA), if intact.

Objective: The investigators aim to study the patient specific threshold for arterial blood pressure to maintain adequate cerebral perfusion (CBFV) in the perioperative setting and the association between perioperative abnormalities with postoperative brain damage and neurobehavioral outcomes.

Study design: In a prospective observational cohort study bilateral cerebral blood flow velocity (CBFV) measurements are performed with transcranial doppler (TCD), together with invasive arterial blood pressure (iABP) measurements in the perioperative period.

Study population: Neonates (semi-) electively scheduled for major cardiac- and non cardiac surgery.

Main study parameters/endpoints: Main study endpoint is the Critical Closing Pressure (CrCP) within and between subjects. Furthermore, we evaluate the association with new white matter injury (WMI) on the postoperative MRI.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Anticipated risks caused by TCD monitoring in neonates are considered negligible when monitoring is executed according to the BMUS guidelines and ALARA principle. Each time energy is converted from one form to another, part of it is inevitably converted to heat. Theoretically, if at all, the maximum temperature rise will happen at the skin- temporal bone side, where the monitoring probes are placed. A maximal thermal index (TI) of 0.7 is allowed, this corresponds with 0.7 o C temperature rise.

Patients might not benefit from participation in this study as the TCD measurements are only visible and available to the TCD operator, and we do not yet know how the results could possibly influence the procedure. However, in the unlikely situation where cerebral perfusion is severely compromised for a longer period of time or in case of occurrence of large air emboli, improper cannulation or cross clamping the cardiac team will be notified. Therefore, a neonate might benefit from participation.

ELIGIBILITY:
Inclusion Criteria:

* Term infant aged < 42 days / Preterm born > 32 weeks and with a corrected age < 42 days
* (Semi-) elective cardiac of major non-cardiac surgery
* Routine placement of an arterial cannula for invasive blood pressure monitoring.

Exclusion Criteria:

* Grade III-IV intracranial hemorrhage.
* Emergency surgery or semi-elective surgery performed out of hours.
* Informed consent from the parents is not obtained.

Max Age: 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible patients are term infants within 42 days (6 weeks) after birth, or infants prematurely born (with a gestational age >32 weeks) at a corrected age of <42 days, who are scheduled for cardiac or non-cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Critical Closing Pressure (CrCP) | During congenital heart surgery
  Detection of the critical closing pressure (CrCP) of the brain, the arterial blood pressure at which brain vessels collapse and cerebral blood flow ceases, in a cohort of neonates who need major cardiac surgery. We hypothesize that neonates have a unique CrCP and cerebral ischemia occurs during episodes with critically endangered blood supply to the brain, when the arterial blood pressure (iABP) is below CrCP.

SECONDARY OUTCOMES:
Incidence white matter injury (WMI) on the postoperative MRI. | Within the first postoperative 10 days
  Compare CrCP between outcome groups, absent or new white matter injury (WMI) on the postoperative MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Kim van Loon, MD, PhD, Principal Investigator — University Medical Center Utrecht / Wilhelmina Children's Hospital
Locations (1):
- UMC Utrecht / Wilhelmina Children's Hospital, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martherus BV, Alderliesten T, Fonteyn EMR, Ceelie I, van Vriesland DJ, Nijman J, Talacua H, Nievelstein RAJ, Dudink J, Benders MJNL, Buhre WFFA, van Loon K. Bilateral Transcranial Doppler Monitoring During Neonatal Cardiac Surgery; Guidance for Clinical and Scientific Use. Paediatr Anaesth. 2025 Dec 24. doi: 10.1002/pan.70106. Online ahead of print. PMID 41439495